CLINICAL TRIAL: NCT02325778
Title: Randomized, Single-blind, Comparative Trial of Two AF Ablation Strategies (CTI Ablation Prior to LA Ablation Versus CTI After LA Ablation) to Eliminate Persistent AF
Brief Title: Comparison of CTI Ablation Prior to or After LA Ablation for AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-01007
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTI First (Experimental): CTI ablation prior to left atrial ablation
  Interventions: Procedure: CTI ablation Timing
- CTI second (Experimental): CTI ablation after left atrial ablation
  Interventions: Procedure: CTI ablation Timing

INTERVENTIONS:
Procedure: CTI ablation Timing — The timing of when the CTI ablation is performed. There are no other relevant interventions used in the procedure.

SUMMARY:
This study is designed to determine if CTI prior to CPVA/PVI/Linear Lesions/Fractionation results in reduced left atrial ablation lesion sets prior to restoration of sinus rhythm in patients with long standing persistent atrial fibrillation in the absence of antiarrhythmic drug therapy compared to CTI after CPVA/PVI/Linear Lesions/Fractionation.

ELIGIBILITY:
Inclusion Criteria:

* continuous/persistent atrial fibrillation

Exclusion Criteria:

* age<18
* congenital heart disease
* pacemaker or ICD implant
* previous ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of Ablation Lines Required to Organize Atrial Fibrillation to an Atrial Tachycardia or Sinus Rhythm | Acute (intra procedure)

SECONDARY OUTCOMES:
Early recurrence of atrial arrhythmias | 3 months
  Atrial Fibrillation or Atrial Tachycardia lasting longer than 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Aizer, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States